CLINICAL TRIAL: NCT05117645
Title: Role of Computed Tomography in Evaluation of Different Causes of Intestinal Obstruction Correlated With Operative Findings
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Alaa Nour Abdelghaffar, resident doctor at radiological and interventional department sohag university hospital, Sohag University
Other Study IDs: soh-med-21-11-04
Record Dates: First submitted 2021-11-10; First posted 2021-11-11 (Actual); Last update posted 2021-11-11 (Actual); Status verified 2021-11

CONDITIONS: Intestinal Obstruction
MeSH Terms: conditions — Intestinal Obstruction | interventions — Tomography, X-Ray Computed

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cases: patients come to surgical emergency unit and complaining of intestinal obstruction and CT Abdomen and pelvis will be done to detect the cause then will be compared with operative findings .
  Interventions: Diagnostic Test: Computed tomography

INTERVENTIONS:
Diagnostic Test: Computed tomography — All patients will be examined by multislice CT scanner,Light speed 5X GE 8 detector elements scanner or GE Revolution Evo 128 multidetector elements scanner (GE Healthcare, Chicago, Illinois, United state) or Toshibe Alexion 16 detector elements scanner (Aplio 500, Toshiba Medical Systems, Otawara-shi, Tochigi 324-8550, Japan). Axial scanns will be done commences at 1 cm above the diaphragm and ending at lesser trochanters then coronal and sagittal reconstruction images will be exposed.

SUMMARY:
Intestinal obstruction is a common clinical problem that occurs secondary to mechanical or functional obstruction of the intestine, preventing normal transit of its contents. It is a frequent cause of hospitalization and represents 15-20% of surgical admissions for acute abdominal pain .

The underlying aetiology of large bowel obstructions (LBOs) is age dependent, but in adulthood, the most common cause is colonic cancer (50-60%), typically in the sigmoid. The second most common cause in adults is acute diverticulitis (involving the sigmoid colon). Together, obstructing tumors and acute diverticulitis account for 90% of all causes of LBO.

Adhesions are the most common cause of small bowel obstruction (SBO) , For practical purposes, they do not tend to cause LBO.Other causes which cause symptoms that are mimic intestinal obstruction as in bowel ischemia that mainly caused by mesenteric vessels occlusion (adynamic obstruction).

Computed tomography (CT) has become a mainstay in diagnosing bowel obstruction. This is because the management of obstruction has dramatically changed with a decrease in the proportion of patients who need surgery Multi Detector Computed Tomography scanners provide a huge gain in performance that can be used to reduce the scan time, reduce section collimation, or to increase scan length surgery.

Diagnosis of intestinal obstruction is established by patient history and clinical findings include abdominal distension, acute abdominal pain, vomiting and inability to pass stools or flatus .

The role of CT in diagnosing intestinal obstruction has been expanding by determining presence, degree, level and cause (extrinsic lesions, intrinsic lesions, intussusception, intraluminal lesions) of obstruction and in identifying any associated strangulation, and also it has an important role in diagnosing the mesenteric vessels obstruction by thrombi by injection of IV contrast media which causes adynamic bowel obstruction .

ELIGIBILITY:
Inclusion Criteria:

* Any age group and gender presented by manifestations of acute intestinal obstruction.

Exclusion Criteria:

* Pregnant women.

Min Age: 1 Year | Sex: Female
Age Groups: Child, Adult, Older Adult
Study Population: patients diagnosed that they have intestinal obstruction of any age group come to surgical emergency unit will be examined by general and local examination then they will be prepared by oral contrast according to their clinical condition , CT abdomen and pelvis will be done and then they will be explored to find out the cause and then results of CT and operative findings will be compared.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-12 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Emphasization the role of the MDCT in the evaluation of intestinal obstruction. | 6 months
  Patients complaining of intestinal obstruction will undergo oral preparation according to their condition then will undergo CT abdomen and pelvis , some of them will undergo exploration others will be observed then comparison with operative findings and observation will be done.

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] van Steensel S, van den Hil LCL, Schreinemacher MHF, Ten Broek RPG, van Goor H, Bouvy ND. Adhesion awareness in 2016: An update of the national survey of surgeons. PLoS One. 2018 Aug 17;13(8):e0202418. doi: 10.1371/journal.pone.0202418. eCollection 2018. PMID 30118503
- [Background] Jaffe T, Thompson WM. Large-Bowel Obstruction in the Adult: Classic Radiographic and CT Findings, Etiology, and Mimics. Radiology. 2015 Jun;275(3):651-63. doi: 10.1148/radiol.2015140916. PMID 25997131
- [Background] De Monti M, Cestaro G, Alkayyali S, Galafassi J, Fasolini F. Gallstone ileus: A possible cause of bowel obstruction in the elderly population. Int J Surg Case Rep. 2018;43:18-20. doi: 10.1016/j.ijscr.2018.01.010. Epub 2018 Feb 4. PMID 29414501